CLINICAL TRIAL: NCT00379015
Title: Neoadjuvant Epirubicin/Cyclophosphamide Followed by Docetaxel Combined With Trastuzumab for the Patients With HER-Positive Advanced Breast Cancer
Brief Title: Epirubicin and Cyclophosphamide Followed By Docetaxel and Trastuzumab in Treating Women With HER2-Positive Stage III or Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000496448; TUSM-BRI-BC04-01
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Cyclophosphamide; Docetaxel; Epirubicin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HER2 over-expressing primary breast cancer group (Experimental): Patients receive epirubicin hydrochloride and cyclophosphamide in week 1-3. Treatment with epirubicin hydrochloride and cyclophosphamide repeats every 3 weeks for 4 courses. Patients then receive docetaxel in week 13 and trastuzumab (Herceptin®) in weeks 13-15. Treatment with docetaxel and trastuzumab repeats every 3 weeks for 4 courses.
  Patients then undergo appropriate surgery. After surgery, patients with hormone receptor-positive disease receive trastuzumab once weekly and either tamoxifen with or without a luteinizing hormone-releasing hormone agonist or an aromatase inhibitor. Treatment continues for 40 weeks.
  Interventions: Biological: trastuzumab; Drug: cyclophosphamide; Drug: docetaxel; Drug: epirubicin hydrochloride; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Biological: trastuzumab
Drug: cyclophosphamide
Drug: docetaxel
Drug: epirubicin hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, cyclophosphamide, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving chemotherapy and a monoclonal antibody before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving epirubicin and cyclophosphamide followed by docetaxel and trastuzumab works in treating women with HER2-positive stage IIIB, stage IIIC, or stage IV primary breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pathological complete response in women with HER2-positive stage IIIB-IV breast cancer treated with neoadjuvant epirubicin hydrochloride and cyclophosphamide followed by docetaxel and trastuzumab (Herceptin®).

Secondary

* Determine the clinical response in patients treated with this regimen.
* Determine the recurrence-free survival of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive epirubicin hydrochloride and cyclophosphamide in weeks 1-3. Treatment with epirubicin hydrochloride and cyclophosphamide repeats every 3 weeks for 4 courses. Patients then receive docetaxel in week 13 and trastuzumab (Herceptin®) in weeks 13-15. Treatment with docetaxel and trastuzumab repeats every 3 weeks for 4 courses.

Patients then undergo appropriate surgery. After surgery, patients with hormone receptor-positive disease receive trastuzumab once weekly and either tamoxifen with or without a luteinizing hormone-releasing hormone agonist or an aromatase inhibitor. Treatment continues for 40 weeks.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary breast cancer

  * Stage IIIB, IIIC, or IV disease
* No inflammatory disease
* HER2 over-expressing tumor as assessed by immunohistochemistry and/or fluorescent in situ hybridization
* Hormone receptor status known

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Performance status 0-1
* WBC ≤ 10,000/mm³
* Absolute neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.5 g/dL
* SGOT/SGPT ≤ 60 IU/L
* Bilirubin ≤ 1.5 mg/dL
* Creatinine ≤ 1.5 mg/dL
* LVEF ≥ 55%
* No signs of pneumonitis

PRIOR CONCURRENT THERAPY:

* No prior surgery except for biopsy
* No prior or concurrent chemotherapy and/or hormonal therapy
* No prior or concurrent biological therapy
* No prior or concurrent radiotherapy except postoperative radiotherapy

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pathological complete response | Whitin the first 7-28 days after the last administration of neoadjuvant therapy of trastuzumab
  Pathological complete response is assessed in surgical resected specimens of primary tumor from patients who underwent a primary radical surgery in this study.

SECONDARY OUTCOMES:
Clinical response | From 7 days after the last adoministration of neosdjuvant therapy of Trastuzumab until surgery.
  Clinical response is assessed as overall response in target lesion of primary tumor from 7 days after the last administration of neoadjuvant therapy of Trastuzumab until surgery.
Pathological response of axillary lymph nodes | Whitin the first 7-28 days after the last administration of neoadjuvant therapy of trastuzumab.
  Pathological response of axillary lymph nodes is assessed in surgical specimens of primary tumor from patients who underwent a primary radical surgery in this study.
Recurrence-free survival | 8 years
  Recurrence-free survival is defined as time from date of enrollment until date of recurrence or death from any cause, whichever comes first.
Overall survival | 8 years
  Overall survival is defined as time from date of enrollment until date of death from any cause.
Adverse event | 70 months
  Types and severities of adverse events from date of starting protocol treatment until 30 days after date of finishing the treatment are evaluated according to Japanese version of the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) by Translational Research Informatics Center.

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Ikeda, MD, Study Chair — Teikyo University
Locations (5):
- Japan (5):
  - Shikoku Cancer Center, Matsuyama, Ehime
  - National Kyushu Cancer Center, Fukuoka, Fukuoka
  - Keio University Hospital, Tokyo, Tokyo
  - Teikyo University School of Medicine, Tokyo, Tokyo
  - Niigata Cancer Center Hospital, Niigata